CLINICAL TRIAL: NCT03280875
Title: Personalisation of Exercise by Muscle Modulation, Step 1: Construction and Validation of an Algorithm for Personalisation for Pedalling Exercises
Brief Title: Creation of an Algorithm for the Personalisation of Pedalling Exercises
Acronym: EXOMODE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Centre Hospitalier Universitaire Dijon (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: Casillas ANR 2015
Record Dates: First submitted 2017-08-04; First posted 2017-09-13 (Actual); Last update posted 2021-07-28 (Actual); Status verified 2021-07

CONDITIONS: Aging

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- healthy volunteers (Experimental)
  Interventions: Other: pedalling exercises

INTERVENTIONS:
Other: pedalling exercises — pedalling exercises on a bicycle ergometer

SUMMARY:
The aim of the EXO-MODE project is to develop an innovative algorithm for the personalisation of Concentric and / or Eccentric training programmes adapted to the individual to improve the efficiency and tolerance. This algorithm will make it possible to personalise trainings programmes according to the different profiles of subjects, determined on the basis of their personal characteristics (age, sex, comorbidities), their exercise capacity and muscle performance, their level of motivation and their perception of the workload, and of the principal objective of the training programme. The final goal is to develop a tool to allow elderly populations to exercise more easily and more effectively.

ELIGIBILITY:
Inclusion Criteria:

* Subject able to understand simple instructions and to provide consent
* Men or women aged 18 to 75 years old.
* Subjects who engage in moderate physical activity (Level 1 or 2 defined by the recommendations for the classification of subjects during performance studies) [2].

Exclusion Criteria:

* Persons without national health insurance cover,
* Cardio-respiratory failure, coronaropathy, severe obstructive cardiomyopathy,
* Recent history of venous thromboembolism (previous 3 months),
* Any medical disorder that could have a major impact on functional capacities (examples: non-stabilised metabolic disorders, such as progressive renal failure, severe asthenia related to a non-stabilised disease, such as neoplasia, systemic disease…),
* Physical disability affecting the lower limbs or the pelvis that could impair or prevent exercise on a cycle ergometer, whether neurological (central or peripheral), arterial (i particular, arteriopathy of the lower limbs with a systolic index < 0.6) or orthopaedic (degenerative or inflammatory rheumatism).
* Pregnant or breast-feeding women

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 133 (Actual)
Dates: Start 2017-05-02 (Actual); Primary Completion 2021-04-28 (Actual); Study Completion 2021-05-13 (Actual)

PRIMARY OUTCOMES:
Preliminary phase: level of perception of effort dissociated from the pain felt | through study phase completion, an average of 3 months
Phase 1:level of pain measured by visual analog scale | through study phase completion, an average of 9 months

CONTACTS AND LOCATIONS:
Locations (1):
- CHU dijon Bourgogne, Dijon, France